CLINICAL TRIAL: NCT07288203
Title: A Phase 2, Multicenter, Open-label Study of Lifileucel (Tumor-infiltrating Lymphocytes [TIL]) in Participants With Previously Treated Advanced Melanoma
Brief Title: A Study of Lifileucel (Tumor-infiltrating Lymphocytes) in Adults With Advanced Melanoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Iovance Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IOV-MEL-202; 2025-522054-40-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-09; First posted 2025-12-17 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Melanoma (Skin Cancer); Unresectable Melanoma; Metastatic Melanoma
Keywords: Tumor Infiltrating Lymphocytes; TIL; Metastatic Melanoma; Unresectable Melanoma; Cell Therapy; Cellular Immuno-therapy; IL-2; Non-myeloablative lymphodepletion (NMALD); Melanoma; Lifileucel; Skin Cancer; LN-144; BRAF v600; BRAF/MEK
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — lifileucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Lifileucel
  Interventions: Biological: Lifileucel

INTERVENTIONS:
Biological: Lifileucel — A tumor sample is resected from each patient for lifileucel manufacturing. Patients will first receive the preparative non-myeloablative lymphodepletion (NMA-LD) regimen. They will then receive the lifileucel infusion, followed by an abbreviated course of aldesleukin.
  Other Names: LN-144

SUMMARY:
This is a Phase 2, multicenter, open-label study of lifileucel (tumor-infiltrating lymphocytes [TIL]) in participants with previously treated advanced melanoma

DETAILED DESCRIPTION:
This is a Phase 2 study of the lifileucel treatment regimen in participants who previously received treatment for unresectable or metastatic (advanced) melanoma with 1 prior line of an anti-programmed cell death protein-1 (PD-1) or anti-programmed death ligand 1 (PD-L1) agent or whose melanoma progressed during and/or within ≤ 12 weeks after adjuvant anti-PD-(L)1 treatment (early relapse). Participants who have BRAF V600 mutation positive melanoma may have received or refused 1 additional prior line treatment with a BRAF inhibitor

± a MEK inhibitor

ELIGIBILITY:
Inclusion Criteria:

* Participant has a histologically or pathologically confirmed diagnosis of Stage IIIC, IIID, or IV unresectable or metastatic melanoma.
* The participant has an ECOG performance status of 0 or 1 and an estimated life expectancy of > 6 months.
* The participant must have experienced radiographic disease progression on: 1 prior line of an anti-PD-(L)1 treatment (as a monotherapy or as part of a combination) for advanced melanoma and/or during or within ≤ 12 weeks after adjuvant anti-PD-(L)1 treatment (as a monotherapy or as part of a combination). Participants who have BRAF V600 mutation positive melanoma may have received 1 additional prior line of treatment with a BRAF inhibitor ± a MEK inhibitor.
* Participant is assessed as having at least one resectable lesion (or aggregate lesions) for lifileucel generation.
* Participant must have at least one measurable disease as defined by RECIST 1.1 following tumor resection.
* Participants who are > 70 years of age may be allowed to enroll after the investigator discusses with the medical monitor.
* Participants of childbearing potential or those with partners of childbearing potential must be willing to practice an approved method of highly effective birth control.
* Participants must have adequate organ function.
* Participant is willing to receive optimal supportive care, including intensive care, from enrollment until the first post-treatment tumor assessment.

Exclusion Criteria:

* Participant has melanoma of uveal/ocular origin.
* Participant has symptomatic untreated brain metastases.
* Participant has active uveitis that requires active treatment.
* Participant has an active medical illness(es) that, in the opinion of the investigator, would pose increased risks for study participation, such as systemic infections; seizure disorders; coagulation disorders; or other active major medical illnesses of the cardiovascular, respiratory, or immune systems.
* Participant has any form of primary or acquired immunodeficiency (eg, SCID or AIDS).
* Participant had another primary malignancy within the previous 3 years (except for those that do not require treatment or were curatively treated >1 year ago, and in the judgment of the investigator do not pose a significant risk of recurrence.)
* Participant has a history of allogeneic cell or organ transplant.
* Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.

Other protocol defined inclusion/exclusion criteria could apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11-28 (Actual); Primary Completion 2032-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 5 years
  To evaluate the efficacy of lifileucel as measured by ORR per RECIST v1.1 as assessed by the IRC

SECONDARY OUTCOMES:
Complete Response Rate | 5 years
  To evaluate the efficacy of lifileucel as measured by CR rate per RECIST v1.1 as assessed by the IRC
Duration of Response | 5 years
  To evaluate the efficacy of lifileucel as measured by DOR per RECIST v1.1 as assessed by the IRC
Disease Control Rate | 5 years
  To evaluate the efficacy of lifileucel as measured by DCR per RECIST v1.1 as assessed by the IRC
Progression-Free Survival | 5 years
  To evaluate the efficacy of lifileucel as measured by PFS per RECIST v1.1 as assessed by the IRC
Objective Response Rate | 5 years
  To evaluate the efficacy of lifileucel as measured by ORR per RECIST v1.1 as assessed by the investigators
Complete Response Rate | 5 years
  To evaluate the efficacy of lifileucel as measured CR rate per RECIST v1.1 as assessed by the investigators
Duration of Response | 5 years
  To evaluate the efficacy of lifileucel as measured by DOR per RECIST v1.1 as assessed by the investigators
Disease Control Rate | 5 years
  To evaluate the efficacy of lifileucel as measured by DCR per RECIST v1.1 as assessed by the investigators
Progression-Free Survival | 5 years
  To evaluate the efficacy of lifileucel as measured by PFS per RECIST v1.1 as assessed by the investigators
Overall Survival | 5 years
  To evaluate the efficacy of lifileucel as measured by OS
Adverse Events | 5 years
  To demonstrate safety and tolerability of lifileucel

CONTACTS AND LOCATIONS:
Locations (5):
- Sarah Cannon Research Institute, Nashville, Tennessee, United States
- Greenslopes Private Hospital, Greenslopes, Queensland, Australia
- Canada (2):
  - Princess Margaret Cancer Centre, Toronto, Ontario, Canada
  - Centre Hospitalier de l'Universite de Montreal, Montral, Quebec, Canada
- Royal Marsden Hospital, London, United Kingdom